CLINICAL TRIAL: NCT06763263
Title: Effect of Superhero Clothing and Figure on Hospital Adjustment in Children During Hospitalization: Randomized Controlled Study
Brief Title: Effect of Superhero Clothing and Figure on Hospital Adjustment in Children During Hospitalization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nisa Meriç Turan (Other)
Responsible Party: Sponsor-Investigator, Nisa Meriç Turan, Master Student/Nurse, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NEUTEZYL2024
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Hospitalization in Children
Keywords: Hospitalization in children; Child; Nursing

STUDY DESIGN:
Intervention Model Description: The study was planned as a pre-test, post-test parallel group (invertion-control), randomized controlled experimental research type.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Superhero Clothing and Figure Group (Experimental): Superhero Clothing and Figure Group
  Interventions: Behavioral: Experimental
- Active:Control (Active Comparator): Control
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Experimental — Children and their parents in this group will be informed about the research and their verbal and written consent will be obtained. A questionnaire will be filled out before the application. Then, the child will be allowed to choose one of the superhero clothes he/she wants in his/her room and will be allowed to wear the clothes. The superhero figure will be shown to him/her and he/she will be allowed to play with the clothes and the figure for 2 hours.
  Arms: Experimental: Superhero Clothing and Figure Group
Behavioral: Control — The children in this group and their parents will be informed about the research and their verbal and written consent will be obtained. A questionnaire will be filled out before the application. The children will be evaluated in terms of their reactions after their hospitalization, they will not be dressed in any clothing and no superhero figures will be used. Then the questionnaire will be filled out again and scoring will be done. In order to prevent ethical bias before discharge, the child will be dressed in a superhero costume and will be allowed to spend time with the clothing and figure.
  Arms: Active:Control

SUMMARY:
Healthcare professionals and administrators who serve children are aware of the role of play in children's lives and with this awareness, they design playrooms and areas for children in hospitals. Nurses who consider play as an important atraumatic care approach that supports the child's development, reduces stress and anxiety, and thus contributes to the improvement of hospital compliance have conducted some studies on this subject. Sarman (2022) found in his study that animal-assisted treatment with aquarium fish in the hospital for children aged 8-10 was effective in reducing children's fear and anxiety, strengthening positive emotions, ensuring that the hospital environment was accepted as safe, reducing the feeling of loneliness and facilitating adaptation to the hospital. In another study, play and art therapy was applied to hospitalized children between the ages of 2 and 4, and it was determined that play therapy was more effective in reducing children's anxiety than art therapy and the control group. In their study evaluating the effect of the "hospital friend, Yarencik" initiative on the hospital adaptation of children aged 1-3, Özcan and Güdücü Tüfekci (2022) found that the hospital adaptation of the intervention group after the application was significantly higher than the control group. Although the above studies show that studies using developmentally appropriate and attractive methods to increase the compliance of young children to hospitalization are effective, the number of methods and studies tested is limited. Finding the best method to increase the compliance of young children to hospital and providing evidence that will form the basis for the development and updating of guides or guides is an important requirement.

DETAILED DESCRIPTION:
Illness and hospitalization are processes that cause negative experiences for the child and the family and that worry and disturb the parents. The number of children affected by chronic diseases or illnesses suffered in the last 6 months in Turkey in 2022 was determined as 6.5%. The illness and hospitalization process affects both the child and the family. In the hospital environment, children can experience many negative emotions such as anxiety, stress, fear, communication problems, anger, regression, hopelessness. Young children, especially those hospitalized, experience adverse psychosocial symptoms. Factors such as the child's gender, age, developmental level, emotional state, parents' level of education and reaction to the disease, level of communication within the family, the child being separated from home or loved ones, whether the disease is acute or chronic, the treatment and adaptation process, feeling pain/suffering, experiencing organ or function loss can affect the child's adaptation to the hospital. Young children may not understand the explanations given about their illness due to their developmental level. Children may experience adaptation problems in the hospital environment with reactions such as fear, anxiety, anger, rage, and thumb sucking.

Parents may also experience psychological or social problems even after their children are hospitalized or discharged. In a study conducted by Açıkgöz et al. (2019) with mothers of 100 hospitalized children diagnosed with acute illness and 100 with chronic illness, 36% of mothers of children with acute illness and 21% of mothers of children with chronic illness had severe depressive symptoms. In the same study, 95% of mothers of children with acute illness had high state anxiety levels, 87% had high trait anxiety levels, and 87% of mothers of children with chronic illness had high state anxiety levels and 69% had high trait anxiety levels. In a study conducted with 118 mothers and fathers whose children were in intensive care, it was found that 24% of the parents had severe anxiety, 51% had major depression and 26% had decisional conflict. The emotions experienced by children, their ability to cope with and adapt to them, and the duration, severity or intensity of the disease affect mothers' concerns.

One of the most important factors that increase the stress or anxiety level of children and families and make adaptation difficult is the traumatizing effect of the child's hospitalization and the events experienced in the hospital environment. In order to reduce these traumatic effects, pediatric nurses apply atraumatic care. Atraumatic care practices include a series of nursing interventions that ensure the active participation of the child and family in care, provision of emotional support, coping with stress, and reduction of pain. Positive experiences during the child's hospitalization period thanks to atraumatic care practices positively affect the child and the family. In this context, many interventions can be made to ensure the child's adaptation to the hospital, such as various games, toys, books, cartoons, videos, family and friend visits, reading books, chatting, writing letters, music activities, painting, theater and clown shows, computer activities, introduction activities and various forms of educational activities, depending on the child's age and development level.

Healthcare professionals and administrators who serve children are aware of the role of play in children's lives and with this awareness, they design playrooms and areas for children in hospitals. Nurses who consider play as an important atraumatic care approach that supports the child's development, reduces stress and anxiety, and thus contributes to the improvement of hospital compliance have conducted some studies on this subject. Sarman (2022) found in his study that animal-assisted treatment with aquarium fish in the hospital for children aged 8-10 was effective in reducing children's fear and anxiety, strengthening positive emotions, ensuring that the hospital environment was accepted as safe, reducing the feeling of loneliness and facilitating adaptation to the hospital. In another study, play and art therapy was applied to hospitalized children between the ages of 2 and 4, and it was determined that play therapy was more effective in reducing children's anxiety than art therapy and the control group. In their study evaluating the effect of the "hospital friend, Yarencik" initiative on the hospital adaptation of children aged 1-3, Özcan and Güdücü Tüfekci (2022) found that the hospital adaptation of the intervention group after the application was significantly higher than the control group. Although the above studies show that studies using developmentally appropriate and attractive methods to increase the compliance of young children to hospitalization are effective, the number of methods and studies tested is limited. Finding the best method to increase the compliance of young children to hospital and providing evidence that will form the basis for the development and updating of guides or guides is an important requirement.

ELIGIBILITY:
Inclusion Criteria:

* The child's age range is between 24-36 months
* On the first day of the child's hospitalization
* The child is hospitalized with an acute problem
* It is the child's first hospitalization
* The child will probably stay in the hospital for at least three days.
* Parent's ability to read and write Turkish
* Parent must be over 18 years of age
* Parent's consent to participate in the research

Exclusion Criteria:

* The child has a mental health problem
* The child receives daily outpatient treatment at the hospital
* Children hospitalized with their siblings
* The parent has a known psychiatric problem
* Parent has communication problems

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic Questionnaire | During the children's first hospitalization, the researcher will fill out Sociodemographic Questionnaire ( Approximately 10 minute).
  This form was prepared by researchers in line with the literature in order to determine the sociodemographic characteristics of the children and to learn their thoughts about the hospital It consists of 14 questions that include the sociodemographic characteristics of the child and the family and information about the hospital.
Children's Hospital Adaptation Evaluation Scale (CHILD-HÜDO) | It will be filled out by the researcher and parent before and after the procedure (Approximately 10 minute).
  The scale, developed in Turkey to evaluate the hospitalization of mothers' 1-3 year old children, is a 5-point Likert-type scale (1-Continuous, 2- Frequently, 3- Occasionally, 4- Very little, 5- Never). It was prepared for children aged 1-3 who are hospitalized. The Scale for Evaluating Children's Hospital Adaptation consists of 22 items and a single dimension. The scale was developed by Özcan and Güdücü Tüfekci by 2022. The lowest score that can be obtained from the scale is 22, and the highest score is 110. As the score obtained from the scale increases, the children's adaptation to the hospital increases. There is no reverse-scored item in the scale. Cronbach's alpha was determined as 0.818 for the entire scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No